CLINICAL TRIAL: NCT03033394
Title: Defining Adult Beta-lactam Antimicrobial Pharmacokinetics Across the Secondary Care Setting
Brief Title: Beta-lactam Pharmacokinetics in Secondary Care
Status: Completed | Type: Observational
Sponsor: Imperial College London (Other)
Responsible Party: Sponsor
Other Study IDs: 207217; 16/LO/2179 (Other: REC); 33017 (Other: NIHR CRN CPMS)
Record Dates: First submitted 2017-01-19; First posted 2017-01-26 (Estimated); Results first posted 2021-08-30 (Actual); Last update posted 2021-08-30 (Actual); Status verified 2021-08

CONDITIONS: Pharmacokinetics; Beta Lactam Adverse Reaction; Penicillin Allergy
Keywords: Penicillins; Drug Monitoring; Pharmacokinetics
MeSH Terms: interventions — Monobactams; Penicillins

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Plasma
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Beta-lactam antibiotic: Observational pharmacokinetic study of non-critical care patients receiving beta-lactam antibiotics for management of infections.
  Interventions: Drug: Beta-lactam antibiotic

INTERVENTIONS:
Drug: Beta-lactam antibiotic — Routine clinical dosing
  Other Names: Penicillin

SUMMARY:
Currently in the UK, TDM is routinely performed for aminoglycosides and glycopeptide antimicrobial agents, given fears over the narrow therapeutic window of these agents and the serious adverse events associated with toxicity. However, in critical care the role of TDM for optimisation of therapy has been demonstrated to help optimise dosing of patients who tend to have variable pharmacokinetic parameters (J. A. Roberts et al,). This is of growing importance given that low concentrations of antimicrobial agents, below a micro-organisms minimum inhibitory concentration (MIC) is believed to be a major driver of AMR. The investigators set out to explore whether similar observations in PK-PD target variability are currently being observed across the secondary care setting (outside of critical care) and whether these appear to be impacting on clinical outcomes.

DETAILED DESCRIPTION:
STUDY PARTICIPANTS

* Participants receiving oral or intravenous therapy will be included in this study.
* Drug level sampling will be undertaken once the participant is at steady state (after at least 5 doses have been administered to those on treatment).
* All patients will be consented using the participation information leaflet and consent form provided in appendix 1.

DRUG LEVEL SAMPLING

* Patients will be identified for inclusion, and researchers will discuss inclusion in the study with the patient and provide clinical information for them to consider. Individuals will be recruited from all areas of secondary care (including, general medicine, general surgery, augmented care, and out-patient parenteral antimicrobial therapy [OPAT]).
* They will then be consented by researchers after being given at least 24 hours to consider this information and as long as the patient has expressed interest in participating to their treating physician.
* This will include permission for basic, anonymised demographic and clinical data to be collected related to the patients infection, for which they are receiving antimicrobial therapy.
* An extra 3mLs of blood will be collected during the patient's routine daily phlebotomy round following their consent. They will be enrolled for up to 72 hours or two days of routine blood tests (whichever is shorter). Up to 10 samples may be taken during the 2 days the patient is enrolled, depending on the number of routine blood tests the patient receives during that day. No more than 3mLs will be taken per each routine blood sample. For example, if the individuals will only have routine blood tests taken at 8am on day 1 and day 2. Then only two extra samples will be taken (3mLs on D1 and 3mLs on D2).
* The time they received their dose of antimicrobials, the length of infusion time (if available), and time the sample was collected will all be recorded.
* PK/PD indices for evaluation will be calculated post-hoc during pharmacokinetic-pharmacodynamic analysis. TDM sampling can occur at any time during the dosing schedule (in line with routine blood testing).
* A standard operating procedure for this study can be found in appendix 3.

SAMPLE PREPARATION AND ANALYSIS

* All blood samples will be allowed to clot and placed on ice. They will be centrifuged at 2,400rpm for 10 minutes. Sera from each sample will be separated into three vials and stored at -80C.
* Beta-lactam concentrations will be measured using validated high-performance liquid chromatography methods.
* Samples will be stored for up to three years post completion of data collection.

  * Consent will be gained for samples to be used for calibration of electrochemical sensors in ex-vivo studies. This will be performed within 90 days of the samples being collected.

PHARMCOKINETIC-PHARMACODYNAMIC MODELLING

* Data will be anonymised and analysed using Pmetrics in R.
* Different pharmacokinetic models will be explored using in built statistical analysis options and visual predictive checks.
* Pharmacodynamic models will then be incorporated into the model using evidence identified in the literature for selection of parameters.
* Monte Carlo simulation will then be used to for simulation of target attainments and analysis of pharmacodynamic outcomes

ELIGIBILITY:
Inclusion Criteria:

* Adult subjects over 18 years old
* Capacity to consent to participation
* Receiving target antimicrobial (amoxicillin, amoxcillin-clavulanate, cefuroxime, ceftriaxone, flucloxacillin, meropenem, piperacillin-tazobactam) for at least 5 doses prior to sampling
* Appropriate venous access (or for venous access to be gained)

Exclusion Criteria:

* Children under 18 years old
* Lacking capacity or prisoner
* Anaemia or bleeding disorder, deemed significant by the patients physician
* Patient's physician deems that they are not suitable for inclusion in the study
* Patients unlikely to be receiving agent for study period

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Participants from a non-critical care setting will be recruited after receiving at least 5 doses of target antimicrobial. Participants receiving oral and intravenous therapy will be eligible.
Sampling Method: Non-Probability Sample
Enrollment: 65 (Actual)
Dates: Start 2017-07-12 (Actual); Primary Completion 2019-08-01 (Actual); Study Completion 2019-08-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Alison H Holmes, MD MPH MBBS, Principal Investigator — Health Protection Research Unit in HCAI & AMR
Locations (1):
- Hammersmith Hospital, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Completed Sampling
Arm/Group | Beta-lactam Antibiotic
Started | 65
Completed | 65
Not Completed | 0
Period: Completed Pharmacokinetic Analysis
Arm/Group | Beta-lactam Antibiotic
Started | 65
Completed | 59
Not Completed | 6
Not completed — Missing data | 1
Not completed — Oral dosing not incorporated into pharmacokinetic model | 3
Not completed — Level taken at incorrect time | 1
Not completed — Pharmacokinetic soffware unable to generate predicted values | 1
Period: Completed Final Analysis
Arm/Group | Beta-lactam Antibiotic
Started | 59
Completed | 58
Not Completed | 1
Not completed — 1 participant excluded from final analysis as an outlier (>1.5 x interquartile range) | 1

BASELINE CHARACTERISTICS:
Arm/Group | Beta-lactam Antibiotic
Number analyzed (Participants) | 65
Age, Categorical [Count of Participants; unit: Participants] — Population: 6 patients excluded from pharmacokinetic analysis:
  * 1 participant missing data
  * 3 oral dosing could not be integrated into model
  * 1 level taken incorrect time
  * 1 model unable to calculate individual predicted value
  Participants
    number analyzed (Participants) | 59
    <=18 years | 0
    Between 18 and 65 years | 32
    >=65 years | 27
Age, Continuous [Median (Inter-Quartile Range); unit: years] — Population: 6 patients excluded from pharmacokinetic analysis:
  * 1 participant missing data
  * 3 oral dosing could not be integrated into model
  * 1 level taken incorrect time
  * 1 model unable to calculate individual predicted value
  years
    number analyzed (Participants) | 59
    (all) | 62 [48 to 72]
Sex: Female, Male [Count of Participants; unit: Participants] — Population: 6 patients excluded from pharmacokinetic analysis:
  * 1 participant missing data
  * 3 oral dosing could not be integrated into model
  * 1 level taken incorrect time
  * 1 model unable to calculate individual predicted value
  Participants
    number analyzed (Participants) | 59
    Female | 18
    Male | 41
Race (NIH/OMB) [Count of Participants; unit: Participants] — Population: 6 patients excluded from pharmacokinetic analysis:
  * 1 participant missing data
  * 3 oral dosing could not be integrated into model
  * 1 level taken incorrect time
  * 1 model unable to calculate individual predicted value
  Participants
    number analyzed (Participants) | 59
    American Indian or Alaska Native | 0
    Asian | 7
    Native Hawaiian or Other Pacific Islander | 0
    Black or African American | 2
    White | 31
    More than one race | 0
    Unknown or Not Reported | 19

OUTCOME MEASURES:

1. Primary Outcome: Fraction of the Dosing Interval Over Which the Concentration of Unbound Drug is Greater Than the Minimum Inhibitory Concentration (fT>MIC)
Description: Minimum inhibitory concentration (MIC) is the concentration required to visibly inhibit microbial growth in vitro. The MIC for each drug was defined by non-species related breakpoints provided in EUCAST v11.0. Results are given as a fraction of the dosing interval over which the concentration of the unbound drug is greater than the MIC.
Time Frame: Two to 10 samples taken during the first 120 hours of antimicrobial therapy
Measure: Median (Inter-Quartile Range); unit: unitless
Groups:
- Amoxicillin; Co-amoxiclav; Ceftriaxone; Flucloxacillin; Meropenem; Piperacillin-tazobactam: Observational pharmacokinetic study of non-critical care patients receiving beta-lactam antibiotics for management of infections.
  Beta-lactam antibiotic: Routine clinical dosing
Arm/Group | Amoxicillin | Co-amoxiclav | Ceftriaxone | Flucloxacillin | Meropenem | Piperacillin-tazobactam
Number analyzed (Participants) | 3 | 7 | 11 | 14 | 13 | 10
unitless | 0.457 [0.417 to 0.479] | 0.429 [0.417 to 0.479] | 0.747 [0.741 to 1.04] | 0.417 [0.285 to 0.700] | 0.333 [0.319 to 0.345] | 1.63 [0.971 to 1.78]

ADVERSE EVENTS:
Time Frame: Mortality outcome collected from time target antimicrobial commenced until time target antimicrobial stopped. This was median 9 days (interquartile range 6-13 days)
Arm/Group | Beta-lactam Antibiotic
All-Cause Mortality (participants affected / at risk) | 1/59
Serious Adverse Events (participants affected / at risk) | 0/59
Other Adverse Events (participants affected / at risk) | 0/59

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol (2018-01-31): https://cdn.clinicaltrials.gov/large-docs/94/NCT03033394/Prot_000.pdf